CLINICAL TRIAL: NCT01072903
Title: The Role of Intestinal Inflammation in the Pathophysiology of IBS
Brief Title: The Role of Intestinal Inflammation in Irritable Bowel Syndrome (IBS)
Acronym: K23
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yehuda Ringel, Associate Professor of Medicine, University of North Carolina, Chapel Hill
Other Study IDs: 08-1106; K23DK075621 (NIH)
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Inflammation; Colon, Irritable; Colonic Diseases, Functional; Irritable Bowel Syndrome
Keywords: inflammation; colon, irritable; Colonic Diseases, Functional; Irritable Bowel Syndrome
MeSH Terms: conditions — Inflammation; Irritable Bowel Syndrome; Colonic Diseases, Functional

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 8 rectosigmoidal intestinal biopsies, stool, and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IBS: Subjects with IBS
- Healthy: Healthy Controls

SUMMARY:
The research project addresses the following hypotheses (A) the normal balance of beneficial and detrimental commensal intestinal bacteria is deranged in IBS, with selective alterations in clinically defined patient subsets i.e., diarrhea predominant IBS (D-IBS) and post-infectious IBS (PI-IBS); (B) these changes in intestinal microflora are associated with sub-clinical mucosal inflammation and activation of the mucosal immune system; and (C) activation of the mucosal immune system leads to alterations in gastrointestinal (GI) functions (i.e., motility and sensation) and functional symptoms.

DETAILED DESCRIPTION:
There are two main aims in the research study. The first aim is to determine whether sub-clinical mucosal inflammation occurs in patients with D-IBS by identifying alterations in mucosal markers for inflammation (inflammatory cytokines and inflammation-related mediators). The second aim is to investigate whether the identifiable alterations in inflammatory markers are associated with specific abnormalities in intestinal motor and sensory functions that are relevant to the pathophysiology of IBS.

ELIGIBILITY:
Inclusion Criteria:

* Any sex, race, or ethnicity.
* At least 18 years of age (no upper age limit).
* D-IBS and M-IBS patients must meet Rome II criteria for IBS and must have been evaluated by a physician to exclude alternative diseases that could explain the symptoms. For the latter, patients' self statement is acceptable (by self-report, no official document is required).
* D-IBS and M-IBS subjects older than 50 years old must have had a colonoscopy in the past 5 years with a normal report. Hemorrhoids, diverticulosis and polyps are allowed.
* Participation in Dr. Whitehead's heterogeneity of IBS research study, or Dr. Ringel's Probiotic Pain Study.

Exclusion Criteria:

* Healthy controls must have no significant or recurring gastrointestinal symptoms.
* Patients and healthy controls should not have a serious, unstable medical condition.
* Patients and healthy controls must have had no gastrointestinal tract surgery other than appendectomy or cholecystectomy, or any abdominal surgery within the past 3 months. Appendectomy and cholecystectomy are allowed if done more than 2 years ago and symptoms were not changed following the surgery.
* Pregnancy and breastfeeding (by self-report).
* No history of inflammatory bowel diseases, celiac disease, or other diagnosis that could explain chronic or recurring bowel symptoms in IBS patients or controls (by self-report).
* Patients and controls should have no history of lactose malabsorption (by self-report).
* Patients and controls should have no history of clinical symptoms of acute infections during the last 8 weeks prior to enrollment in the study.
* Patients and controls should have no history of anti-inflammatory agents including aspirin, non-aspirin, non-steroid anti-inflammatory (NSAID), steroids, antibiotic, or probiotics treatment during the last 4 weeks prior to enrollment in the study.
* Patients should not have an implanted or portable electro-mechanical medical device such as a pacemaker and/or other implanted stimulators or pumps.
* Evidence of acute inflammation on routine histology.
* Evidence of enteric pathogens on routine stool cultures.
* Presence of a medical condition that requires routine use of antibiotic treatment with dental or other invasive procedures (by self-report).
* To be confirmed at time of screening and the week of the flexible sigmoidoscopy appointment for IBS-M subjects ONLY: In the past week, subject cannot have less than 3 (0-2) bowel movements. Also, in the past week, subject cannot have hard/lumpy stools for 2 or more days.

Only subjects with IBS may participate in the optional SmartPill testing. Subjects are excluded from SmartPill testing if a subject has:

* A history of gastric bezoar.
* Suspected strictures, fistulas, colon cancer or other physiological GI obstruction.
* Dysphagia.
* Diverticulitis.
* Tobacco use within eight hours prior to capsule ingestion and during the initial 8 hour recording on Day 0 or the Ingestion visit.
* Alcohol use within eight hours prior to capsule ingestion and throughout the entire monitoring period (5 days).
* Body Mass Index > 40 kg/m2.
* Female of childbearing age who is not practicing birth control and/or are pregnant or lactating.
* Cardiovascular, endocrine, renal, or other chronic disease likely to affect motility.
* A medical device such as a pacemaker, infusion pump, or insulin pump.
* Any contraindication to use of Fleets Enema or the balloon expulsion test.
* Uncontrolled diabetes with a hemoglobin A1C greater than 10.
* Allergies to any of the ingredients of the standard SmartBar meal
* Subject plans to take any of the following prohibited medications: Medication to alter gastric pH, Medication that affect GI motility for 3 full days before the start of the study and during the ensuing days of study, Medication for nausea and vomiting that block serotonin receptors, Anti-diarrheal agents, Opiate agents used to treat diarrhea, Non-steroidal anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research plans to study 33 diarrhea predominant Irritable Bowel Syndrome and IBS-mixed/alternators patients with current symptom activity (abdominal pain at least once a week in the past month) and 33 healthy controls. The subjects will be of any gender, race or ethnicity and at least 18 years of age. Recruitment for the proposed study takes advantage of an ongoing NIH-supported research study on the heterogeneity of IBS (NIDDK Grant DK 31369, WE Whitehead - PI, IRB#01-1397, GCRC# 1846) currently conducted at UNC.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ringel, MD, Principal Investigator — UNC Chapel Hill Department of Gastroenterology and Hepatology
Locations (1):
- University of North Carolina at Chapel Hill, Program in Digestive Health and the Department of Gastroenterology and Hepatology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Ringel Y, Carroll IM. Alterations in the intestinal microbiota and functional bowel symptoms. Gastrointest Endosc Clin N Am. 2009 Jan;19(1):141-50, vii. doi: 10.1016/j.giec.2008.12.004. PMID 19232285
- [Background] Ringel Y, Drossman DA. Irritable bowel syndrome: classification and conceptualization. J Clin Gastroenterol. 2002 Jul;35(1 Suppl):S7-10. doi: 10.1097/00004836-200207001-00003. PMID 12184143